CLINICAL TRIAL: NCT06268977
Title: Efficacy and Safety of Incorporating Sodium-glucose Cotransporter-2 Inhibitors to Regimens of Diabetes Patients Already Receiving Therapy
Brief Title: Using of SGLt2 Inhibitors in Patients With Type 2 DM
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Caroline Refaat labib, Resident doctor, Assiut University
Other Study IDs: SGLt2i in diabetic type 2
Record Dates: First submitted 2024-01-17; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: SGLT2 inhibitor — a class of prescription medicines that are FDA-approved for use with diet and exercise to lower blood sugar in adults with type 2 diabetes.
  Other Names: gliflozins or flozins

SUMMARY:
To detect the efficacy of SGLT2i in improving the metabolic parameters in patients with type 2 diabetes.

- To detect the side-effects of SGLT2i

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2DM) is a worldwide health problem, with a continuously increasing prevalence . Good management of blood glucose level is critical to delay progression of the underlying metabolic dysfunction and to reduce the risk of diabetic complications . Sodium-glucose cotransporter-2 inhibitors (SGLT2i) are a new class of antidiabetic drug acting by increasing urinary glucose excretion. First approved in 2014, SGLT2i have been widely used to treat patients with type 2 diabetes They are effective in reducing blood glucose, and surprisingly have shown benefits beyond glycaemic control .

Physicians have reported improved hypertension, heart failure, chronic kidney disease, fatty liver disease and obesity However, SGLT inhibitors are not magical drugs, and their use is not free of side effects ( Reported side effects include urinary tract infections, genital infection, dehydration, and hypotension, plus the usual side effects of antidiabetic medications as hypoglycemia . The optimum practical guideline for adding SGLT2 inhibitors to treatment regimens of patients with diabetes is controversial .Many local guidelines and treatment policies exist, yet we need to develop our own local policy at Assiut University hospitals to suit our patients needs and expectations, balancing between efficacy and side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥18 years)
2. both genders ( male and female)
3. type 2 diabetic patients

Exclusion Criteria:

1. history of svere hypoglycemia
2. patients with history of weight loss
3. Patients with history of recurrent UTI

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult diabetic type 2patients
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Effect of adding SGLTi on BP | Six months
  Compare the effect on blood pressure measurement ( SBP and DBP in mmHg) in SGLTi receivers and non SGLTi receivers
Effect of adding SGLTi on BMI | Six months
  compare the effect on BMI ( weight in kg and height in m2) in SGLTi receivers and non SGLTi receivers.

REFERENCES:
- [Background] Sun H, Saeedi P, Karuranga S, Pinkepank M, Ogurtsova K, Duncan BB, Stein C, Basit A, Chan JCN, Mbanya JC, Pavkov ME, Ramachandaran A, Wild SH, James S, Herman WH, Zhang P, Bommer C, Kuo S, Boyko EJ, Magliano DJ. IDF Diabetes Atlas: Global, regional and country-level diabetes prevalence estimates for 2021 and projections for 2045. Diabetes Res Clin Pract. 2022 Jan;183:109119. doi: 10.1016/j.diabres.2021.109119. Epub 2021 Dec 6. PMID 34879977
- [Background] Levine MJ. Empagliflozin for Type 2 Diabetes Mellitus: An Overview of Phase 3 Clinical Trials. Curr Diabetes Rev. 2017;13(4):405-423. doi: 10.2174/1573399812666160613113556. PMID 27296042
- [Background] Vukadinovic D, Abdin A, Anker SD, Rosano GMC, Mahfoud F, Packer M, Butler J, Bohm M. Side effects and treatment initiation barriers of sodium-glucose cotransporter 2 inhibitors in heart failure: a systematic review and meta-analysis. Eur J Heart Fail. 2022 Sep;24(9):1625-1632. doi: 10.1002/ejhf.2584. Epub 2022 Jul 8. PMID 35730422